CLINICAL TRIAL: NCT01184105
Title: A Phase I, Single-Center, Double-Blind, Randomized, Placebo-Controlled, Safety and Pharmacokinetic Study to Evaluate Systemic and Local Vaginal Exposure to Lidocaine and Prilocaine and the Metabolites, 2,6-Dimethylaniline (2,6-DMA) and O-Toluidine, in Female Healthy Volunteer Subjects Following Daily Application of 60 mg PSD502 or Placebo to the Vagina and Cervix for 7 Days
Brief Title: A Safety and Tolerability of PSD502 (a Topical Anesthetic) in the Treatment of Premature Ejaculation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Plethora Solutions Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSD502-PE-007
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2015-09

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (pre) (Experimental): Active treatment or placebo
  Interventions: Drug: Intervention A; Drug: Intervention B
- Cohort 2 (post) (Experimental): Active treatment or placebo
  Interventions: Drug: Intervention A; Drug: Intervention B

INTERVENTIONS:
Drug: Intervention A — A single dose of 60 mg will consist of 6 sprays of the 10 mg strength spray applied topically to cervix (2 sprays) and vaginal fornices (4 sprays)
Drug: Intervention B — A dose of placebo will consist of 6 sprays of the placebo spray applied topically to cervix (2 sprays) and vaginal fornices (4 sprays)

SUMMARY:
A phase I, single-center, double-blind, randomized, placebo-controlled, safety and pharmacokinetic study to evaluate systemic and local vaginal exposure to lidocaine and prilocaine and the metabolites, 2,6-dimethylaniline (2,6-DMA) and o-toluidine, in female healthy volunteer subjects following daily application of 60 mg PSD502 or placebo to the vagina and cervix for seven days

DETAILED DESCRIPTION:
The study drug is a metered-dose anesthetic spray, which is being developed for the treatment of premature ejaculation (PE). The use of anesthetic in topical creams has been well established. The use of a cream does not result in the concentrated drug being in direct contact with the cells, unlike the spray.

Seven clinical studies have already been carried out for the spray in the development of PE. These studies have demonstrated a prolongation of intravaginal ejaculatory latency time and no safety concerns for male patients or their female partners. The partners of clinical study participants have been asked to report health changes during the studies. Reports of vaginal numbness were uncommon; however, effects of the transfer to a partner cannot be excluded. This study is being conducted to investigate in detail the systemic exposure to PSD502 spray in order to assess safety in the female partner. The dose level has been chosen because the total dose applied to the male glans penis is 30 mg, and thus it is potentially possible that his partner could be exposed to this dose. Therefore, the 60 mg dose was chosen to provide safety information with a higher margin of exposure.

ELIGIBILITY:
Inclusion Criteria:

* Female non-smokers aged 18 years old and over
* Willing and able to provide written informed consent
* Generally, in good health in the opinion of the investigator
* Subject must have a body mass index between 18 and 30 kg/m2, inclusive
* Willing and able to comply with all study procedures in the opinion of the investigator
* Negative Papanicolaou (Pap) smear performed during gynecological examination at screening (i.e., Pap smear result that reads negative for any intraepithelial lesions and reparative or reactive changes and with no sign or presence of infection [e.g., bacterial vaginosis, candida, bacterial flora, etc])
* Negative drugs of abuse and cotinine test at screening
* Female subjects of child-bearing potential who are sexually active or become sexually active must be using a method of effective contraception from 14 days before screening and continue to use until the end of the study. If oral contraceptives are used, these must have been stable for a period of 3 months. If a barrier method is being used, this should be latex based and not polyurethane based
* Female subjects who are post-menopausal must have been post-menopausal >1 year and have confirmed elevated serum follicle stimulating hormone at screening

Exclusion Criteria:

* History of a significant medical condition that would preclude further study participation in the opinion of the investigator
* Currently taking, or has taken within the 2 weeks prior to screening, any concomitant medication that could confound interpretation of the safety or pharmacokinetic data on PSD502. Use of prescription medication within 14 days or over-the-counter products within 7 days prior to first dose
* Suffering from a sexually transmitted disease, or is positive for hepatitis B, hepatitis C, human papillomavirus, or human immunodeficiency virus infection
* Safety testing: abnormalities at screening, in particular liver function tests, that are indicative of a medical condition and that would preclude further participation in the opinion of the investigator
* Significant abnormality of the vaginal mucosa or cervix that would preclude interpretation of the examination of these areas or that could be worsened by use of PSD502
* History of alcohol or drug abuse within 1 year prior to screening
* Known drug sensitivity to amide-type local anesthetics
* Unlikely to understand or be able to comply with study procedures, for any reason, in the opinion of the investigator
* History of glucose-6-phosphate dehydrogenase deficiency or use of medications that would increase susceptibility to methemoglobinemia (e.g., anti-malarial agents)
* Use of class I (e.g., mexiletine, tocainide) and III (e.g., amiodarone, sotalol) anti-arrhythmic drugs
* Subject has received an investigational (non-registered) drug within 60 days of screening
* Subjects having any physical or psychological condition that would prevent them from undertaking the study procedures, including but not limited to, the following:

  * Uro-gynecological disease or recent genito-urinary surgery within 8 weeks of screening which would make intravaginal application or vaginal examination/colposcopy difficult or painful or
  * Ongoing significant psychiatric disorder (e.g., bipolar disease, depression/anxiety disorder or schizophrenia)
* Subject has a clinically obvious vaginal infection, such as active vaginal Candida albicans (thrush), or other abnormal vaginal discharge
* Subjects who are pregnant or lactating
* Subjects should not be menstruating during the treatment phase
* Donation of blood or blood products within 60 days prior to dosing or at any time during the study, except as required by this protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety of repeated application of PSD502 to the cervix and vaginal fornices in healthy female subjects. | Days 1 to 7
  Safety assessments consists of monitoring and recording of all adverse events and vital signs, electrocardiograms, physical examinations, and clinical laboratory tests

SECONDARY OUTCOMES:
Extent of systemic absorption of the active ingredients and their metabolites was determined by pharmacokinetic parameters | Days 1 to 7
  Pharmacokinetic parameters: AUC0-t, AUC0-inf, AUCtau, Rc, Cmax, tmax, t½ and kel

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi